CLINICAL TRIAL: NCT04398316
Title: High Dose Intravenous Lidocaine vs Hydromorphone for Acute Abdominal Pain in the Emergency Department: A Randomized, Comparative Efficacy Trial
Brief Title: High Dose IV Lidocaine vs Hydromorphone for Abdominal Pain in the Emergency Department
Acronym: HIDO-LIDO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20202020
Record Dates: First submitted 2020-05-07; First posted 2020-05-21 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Abdominal Pain; Renal Colic
Keywords: lidocaine; hydromorphone; abdominal pain
MeSH Terms: conditions — Abdominal Pain; Renal Colic | interventions — Lidocaine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Lidocaine (Experimental): Administered at a dose of 2 mg/kg over 5 minutes
  Interventions: Drug: Lidocaine Iv
- Intravenous Hydromorphone (Active Comparator): Administered at a dose of 1 mg over 5 minutes
  Interventions: Drug: HYDROmorphone Injection

INTERVENTIONS:
Drug: Lidocaine Iv — 2 mg/kg over 5 minutes
  Other Names: Xylocaine
  Arms: Intravenous Lidocaine
Drug: HYDROmorphone Injection — 1 mg over 5 minutes
  Other Names: Dilaudid
  Arms: Intravenous Hydromorphone

SUMMARY:
Intravenous lidocaine will be given at a dose of 2 mg/kg intravenously to patients in the emergency department with a diagnosis of acute abdominal pain. Its efficacy will be compared to 1 mg of intravenous hydromorphone, with a primary endpoint of mean improvement of pain at 90 minutes.

DETAILED DESCRIPTION:
Abdominal pain is a common chief complaint for patients presenting to the emergency department (ED) in the United States. Intravenous opioids are commonly used to treat acute abdominal pain in the ED. These medications are highly efficacious and, when used in a monitored setting such as the ED, extremely safe. Use of opioids has fallen out of favor because of a spike in opioid-related overdose deaths throughout the United States. While use of opioids in the ED is unlikely to contribute to outpatient opioid deaths, minimizing the use of opioids in the ED will contribute to an opioid free culture, in which opioids are used only when absolutely necessary. A variety of different types of medications can be used in lieu of opioids. One such medication, intravenous lidocaine, has been used extensively for neuropathic pain, in the peri- and post-operative surgical setting, the cardiac care unit, and most recently in the emergency department.

Intravenous lidocaine has long been used to treat pain. In publications dating back to 1980, intravenous lidocaine has been shown to be an effective treatment for neuropathic pain. In the postoperative setting, intravenous lidocaine decreased pain and decreased the need for opiates. More recently, emergency medicine investigators in Iran demonstrated that intravenous lidocaine decreased pain associated with renal colic and limb ischemia. An ED-based study in the United States showed comparable efficacy between morphine and intravenous lidocaine when used for acute pain. Most recently, a prospective RCT showed 120 mg of intravenous lidocaine was efficacious for abdominal pain, albeit not as effective as 1 mg of hydromorphone. However, a subgroup analysis showed that when lidocaine was dosed at 2 mg/kg, it was equally as effective as hydromorphone.

Over the years, intravenous lidocaine has been used for a variety of indications including arrhythmia prophylaxis in patients with acute coronary syndromes. Known side effects of intravenous lidocaine range from transient neurological symptoms (dizziness, paresthesias), to cardiac dysrhythmias and seizure. To date, no deaths have been attributed to its use for treating pain, and the only documented significant complication was due to an unintentional overdose when a patient received ten times the normal dose. All reported side effects in pain patients have been transient and resolved by either stopping the drug, decreasing the infusion rate or by observation alone. Additionally, doses of 2 mg/kg have been tolerated well in the outpatient setting, operating room and ED without any serious side effects. Thus, intravenous lidocaine is an emerging medication for safe and rapid relief of pain, has no known addictive properties, and creates a potential for a pain practice paradigm shift in the United States.

We therefore propose a randomized, double blind, comparative efficacy trial to address the following aim:

To determine if a 2 mg/kg dose of intravenous lidocaine is as equally efficacious as a single dose of 1 mg intravenous hydromorphone for acute abdominal pain in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient in the emergency department (ED)
* Must have acute abdominal pain, defined as abdominal or flank pain of a duration of 7 days or less
* Predicted treatment must include the use of an intravenous opiate

Exclusion Criteria:

* Cardiac conduction system impairment (QTc duration > 0.5s, QRS duration > 0.12s, PR interval <0.12s or > 0.2s)
* Known renal (CKD >2) or liver disease (Childs-Pugh B or greater)
* Hemodynamically instability, defined by the attending physician
* Pregnant or breastfeeding
* Have a known allergy to either medication
* Used of prescription or illicit opioids within the previous week
* Patients with a chronic pain disorder, defined as use of any analgesic medication on more days than not during the four weeks preceding the acute episode of pain

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Chinn, DO, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tremont-Lukats IW, Challapalli V, McNicol ED, Lau J, Carr DB. Systemic administration of local anesthetics to relieve neuropathic pain: a systematic review and meta-analysis. Anesth Analg. 2005 Dec;101(6):1738-1749. doi: 10.1213/01.ANE.0000186348.86792.38. PMID 16301253
- [Background] Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Weibel S. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Database Syst Rev. 2015 Jul 16;(7):CD009642. doi: 10.1002/14651858.CD009642.pub2. PMID 26184397
- [Background] Ventham NT, Kennedy ED, Brady RR, Paterson HM, Speake D, Foo I, Fearon KC. Efficacy of Intravenous Lidocaine for Postoperative Analgesia Following Laparoscopic Surgery: A Meta-Analysis. World J Surg. 2015 Sep;39(9):2220-34. doi: 10.1007/s00268-015-3105-6. PMID 26044546
- [Background] Sun Y, Li T, Wang N, Yun Y, Gan TJ. Perioperative systemic lidocaine for postoperative analgesia and recovery after abdominal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2012 Nov;55(11):1183-94. doi: 10.1097/DCR.0b013e318259bcd8. PMID 23044681
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Background] Marret E, Rolin M, Beaussier M, Bonnet F. Meta-analysis of intravenous lidocaine and postoperative recovery after abdominal surgery. Br J Surg. 2008 Nov;95(11):1331-8. doi: 10.1002/bjs.6375. PMID 18844267
- [Background] Fitzpatrick BM, Mullins ME. Intravenous lidocaine for the treatment of acute pain in the emergency department. Clin Exp Emerg Med. 2016 Jun 30;3(2):105-108. doi: 10.15441/ceem.15.103. eCollection 2016 Jun. PMID 27752626
- [Background] Soleimanpour H, Hassanzadeh K, Mohammadi DA, Vaezi H, Esfanjani RM. Parenteral lidocaine for treatment of intractable renal colic: a case series. J Med Case Rep. 2011 Jun 29;5:256. doi: 10.1186/1752-1947-5-256. PMID 21714904
- [Background] Soleimanpour H, Hassanzadeh K, Vaezi H, Golzari SE, Esfanjani RM, Soleimanpour M. Effectiveness of intravenous lidocaine versus intravenous morphine for patients with renal colic in the emergency department. BMC Urol. 2012 May 4;12:13. doi: 10.1186/1471-2490-12-13. PMID 22559856
- [Background] Firouzian A, Alipour A, Rashidian Dezfouli H, Zamani Kiasari A, Gholipour Baradari A, Emami Zeydi A, Amini Ahidashti H, Montazami M, Hosseininejad SM, Yazdani Kochuei F. Does lidocaine as an adjuvant to morphine improve pain relief in patients presenting to the ED with acute renal colic? A double-blind, randomized controlled trial. Am J Emerg Med. 2016 Mar;34(3):443-8. doi: 10.1016/j.ajem.2015.11.062. Epub 2015 Dec 1. PMID 26704774
- [Background] Vahidi E, Shakoor D, Aghaie Meybodi M, Saeedi M. Comparison of intravenous lidocaine versus morphine in alleviating pain in patients with critical limb ischaemia. Emerg Med J. 2015 Jul;32(7):516-9. doi: 10.1136/emermed-2014-203944. Epub 2014 Aug 21. PMID 25147364
- [Background] Clattenburg EJ, Nguyen A, Yoo T, Flores S, Hailozian C, Louie D, Herring AA. Intravenous Lidocaine Provides Similar Analgesia to Intravenous Morphine for Undifferentiated Severe Pain in the Emergency Department: A Pilot, Unblinded Randomized Controlled Trial. Pain Med. 2019 Apr 1;20(4):834-839. doi: 10.1093/pm/pny031. PMID 29741660
- [Background] Chinn E, Friedman BW, Naeem F, Irizarry E, Afrifa F, Zias E, Jones MP, Pearlman S, Chertoff A, Wollowitz A, Gallagher EJ. Randomized Trial of Intravenous Lidocaine Versus Hydromorphone for Acute Abdominal Pain in the Emergency Department. Ann Emerg Med. 2019 Aug;74(2):233-240. doi: 10.1016/j.annemergmed.2019.01.021. Epub 2019 Feb 26. PMID 30819520
- See also: Emergency Department Visits for Chest Pain and Abdominal Pain: United States, 1999-2008 — https://www.cdc.gov/nchs/data/databriefs/db43.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.33 (13.58) | 61 (0) | 43.25 (16.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White (Caucasian, Non-Hispanic) | 1 | 1 | 2
  Race: Black (African American or African) | 1 | 0 | 1
  Race: American Indian (Native American) or Alaskan Native | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Improvement in Pain at 90 Minutes
Description: The difference between the pain score at time 0 and 90 minutes. Pain score ranges from 0 (no pain) to 10 (maximum pain).
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
score on a scale | 3.67 (3.51) | -1 (0)

2. Secondary Outcome: Sufficient Pain Relief
Description: Does the patient require off-protocol medication for additional pain relief? Off-protocol defined as any opiate or NSAID
Time Frame: From administration of study drug until patient leaves the emergency department, up until 3 hours from administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
Participants | 2 | 1

3. Secondary Outcome: Improvement in Numerical Pain Score at 15 Minutes
Description: The difference between the pain score at time 0 and 15 minutes. Pain score ranges from 0 (no pain) to 10 (maximum pain).
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
score on a scale | 4.33 (3.51) | 0 (0)

4. Secondary Outcome: Improvement in Numerical Pain Score at 30 Minutes
Description: The difference between the pain score at time 0 and 30 minutes. Pain score ranges from 0 (no pain) to 10 (maximum pain).
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
score on a scale | 2.33 (1.53) | 1 (0)

5. Secondary Outcome: Improvement in Numerical Pain Score at 60 Minutes
Description: The difference between the pain score at time 0 and 60 minutes. Pain score ranges from 0 (no pain) to 10 (maximum pain).
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
score on a scale | 4 (3) | 1 (0)

6. Secondary Outcome: Improvement in Numerical Pain Score at 120 Minutes
Description: The difference between the pain score at time 0 and 120 minutes. Pain score ranges from 0 (no pain) to 10 (maximum pain).
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
score on a scale | 4 (3) | -2 (0)

7. Secondary Outcome: Improvement in Numerical Pain Score at 150 Minutes
Description: The difference between the pain score at time 0 and 150 minutes. Pain score ranges from 0 (no pain) to 10 (maximum pain).
Time Frame: 150 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
score on a scale | 3.33 (2.08) | -2 (0)

8. Secondary Outcome: Improvement in Numerical Pain Score at 180 Minutes
Description: The difference between the pain score at time 0 and 180 minutes. Pain score ranges from 0 (no pain) to 10 (maximum pain).
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
score on a scale | 3.33 (2.08) | -2 (0)

9. Secondary Outcome: Patient Preference for the Medication They Received
Description: If the patient were to come to the ED again for the same complaint, would they want the same study drug they received?
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
Participants | 1 | 1

10. Secondary Outcome: Side Effects
Description: Yes or no, did the patient have any side effects, defined as any new symptom after the administration of the study drug.
Time Frame: 15 minutes after administration of study drug then again at 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes and at 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
Participants
  15 Minutes: None | 2 | 1
  15 Minutes: Nausea | 0 | 0
  15 Minutes: Vomiting | 0 | 0
  15 Minutes: Dizziness | 0 | 0
  15 Minutes: Lightheadedness | 0 | 0
  15 Minutes: Paresthesia | 0 | 0
  15 Minutes: Weakness | 0 | 0
  15 Minutes: Slurred speech | 0 | 0
  15 Minutes: Feeling tired | 0 | 0
  15 Minutes: Headache | 1 | 0
  15 Minutes: Other | 0 | 0
  30 Minutes: None | 2 | 1
  30 Minutes: Nausea | 0 | 0
  30 Minutes: Vomiting | 0 | 0
  30 Minutes: Dizziness | 0 | 0
  30 Minutes: Lightheadedness | 0 | 0
  30 Minutes: Paresthesia | 0 | 0
  30 Minutes: Weakness | 0 | 0
  30 Minutes: Slurred speech | 0 | 0
  30 Minutes: Feeling tired | 0 | 0
  30 Minutes: Headache | 1 | 0
  30 Minutes: Other | 0 | 0
  60 Minutes: None | 1 | 1
  60 Minutes: Nausea | 0 | 0
  60 Minutes: Vomiting | 0 | 0
  60 Minutes: Dizziness | 0 | 0
  60 Minutes: Lightheadedness | 0 | 0
  60 Minutes: Paresthesia | 0 | 0
  60 Minutes: Weakness | 0 | 0
  60 Minutes: Slurred speech | 0 | 0
  60 Minutes: Feeling tired | 1 | 0
  60 Minutes: Headache | 1 | 0
  60 Minutes: Other | 0 | 0
  90 Minutes: None | 1 | 1
  90 Minutes: Nausea | 1 | 0
  90 Minutes: Vomiting | 0 | 0
  90 Minutes: Dizziness | 0 | 0
  90 Minutes: Lightheadedness | 0 | 0
  90 Minutes: Paresthesia | 1 | 0
  90 Minutes: Weakness | 0 | 0
  90 Minutes: Slurred speech | 0 | 0
  90 Minutes: Feeling tired | 0 | 0
  90 Minutes: Headache | 0 | 0
  90 Minutes: Other | 0 | 0
  120 Minutes: None | 3 | 1
  120 Minutes: Nausea | 0 | 0
  120 Minutes: Vomiting | 0 | 0
  120 Minutes: Dizziness | 0 | 0
  120 Minutes: Lightheadedness | 0 | 0
  120 Minutes: Paresthesia | 0 | 0
  120 Minutes: Weakness | 0 | 0
  120 Minutes: Slurred speech | 0 | 0
  120 Minutes: Feeling tired | 0 | 0
  120 Minutes: Headache | 0 | 0
  120 Minutes: Other | 0 | 0
  150 Minutes: None | 3 | 1
  150 Minutes: Nausea | 0 | 0
  150 Minutes: Vomiting | 0 | 0
  150 Minutes: Dizziness | 0 | 0
  150 Minutes: Lightheadedness | 0 | 0
  150 Minutes: Paresthesia | 0 | 0
  150 Minutes: Weakness | 0 | 0
  150 Minutes: Slurred speech | 0 | 0
  150 Minutes: Feeling tired | 0 | 0
  150 Minutes: Headache | 0 | 0
  150 Minutes: Other | 0 | 0
  180 Minutes: None | 3 | 1
  180 Minutes: Nausea | 0 | 0
  180 Minutes: Vomiting | 0 | 0
  180 Minutes: Dizziness | 0 | 0
  180 Minutes: Lightheadedness | 0 | 0
  180 Minutes: Paresthesia | 0 | 0
  180 Minutes: Weakness | 0 | 0
  180 Minutes: Slurred speech | 0 | 0
  180 Minutes: Feeling tired | 0 | 0
  180 Minutes: Headache | 0 | 0
  180 Minutes: Other | 0 | 0
  7 Days: None | 3 | 0
  7 Days: Nausea | 0 | 1
  7 Days: Vomiting | 0 | 0
  7 Days: Dizziness | 0 | 0
  7 Days: Lightheadedness | 0 | 0
  7 Days: Paresthesia | 0 | 0
  7 Days: Weakness | 0 | 0
  7 Days: Slurred speech | 0 | 0
  7 Days: Feeling tired | 0 | 0
  7 Days: Headache | 0 | 0
  7 Days: Other | 0 | 0

11. Secondary Outcome: Medication for Side Effects
Description: Are any medications required to control medication side effects, defined as any new symptom after the administration of the study drug?
Time Frame: 15 minutes after administration of study drug then again at 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes and 180 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
Participants
  15 Minutes: None | 3 | 1
  15 Minutes: Diphenhydramine | 0 | 0
  15 Minutes: Ondansetron | 0 | 0
  15 Minutes: Metoclopramide | 0 | 0
  15 Minutes: Droperidol | 0 | 0
  15 Minutes: Promethazine | 0 | 0
  15 Minutes: Prochlorperazine | 0 | 0
  15 Minutes: Other | 0 | 0
  30 Minutes: None | 3 | 1
  30 Minutes: Diphenhydramine | 0 | 0
  30 Minutes: Ondansetron | 0 | 0
  30 Minutes: Metoclopramide | 0 | 0
  30 Minutes: Droperidol | 0 | 0
  30 Minutes: Promethazine | 0 | 0
  30 Minutes: Prochlorperazine | 0 | 0
  30 Minutes: Other | 0 | 0
  60 Minutes: None | 3 | 1
  60 Minutes: Diphenhydramine | 0 | 0
  60 Minutes: Ondansetron | 0 | 0
  60 Minutes: Metoclopramide | 0 | 0
  60 Minutes: Droperidol | 0 | 0
  60 Minutes: Promethazine | 0 | 0
  60 Minutes: Prochlorperazine | 0 | 0
  60 Minutes: Other | 0 | 0
  90 Minutes: None | 2 | 1
  90 Minutes: Diphenhydramine | 1 | 0
  90 Minutes: Ondansetron | 0 | 0
  90 Minutes: Metoclopramide | 0 | 0
  90 Minutes: Droperidol | 0 | 0
  90 Minutes: Promethazine | 0 | 0
  90 Minutes: Prochlorperazine | 0 | 0
  90 Minutes: Other | 0 | 0
  120 Minutes: None | 3 | 1
  120 Minutes: Diphenhydramine | 0 | 0
  120 Minutes: Ondansetron | 0 | 0
  120 Minutes: Metoclopramide | 0 | 0
  120 Minutes: Droperidol | 0 | 0
  120 Minutes: Promethazine | 0 | 0
  120 Minutes: Prochlorperazine | 0 | 0
  120 Minutes: Other | 0 | 0
  150 Minutes: None | 3 | 1
  150 Minutes: Diphenhydramine | 0 | 0
  150 Minutes: Ondansetron | 0 | 0
  150 Minutes: Metoclopramide | 0 | 0
  150 Minutes: Droperidol | 0 | 0
  150 Minutes: Promethazine | 0 | 0
  150 Minutes: Prochlorperazine | 0 | 0
  150 Minutes: Other | 0 | 0
  180 Minutes: None | 3 | 1
  180 Minutes: Diphenhydramine | 0 | 0
  180 Minutes: Ondansetron | 0 | 0
  180 Minutes: Metoclopramide | 0 | 0
  180 Minutes: Droperidol | 0 | 0
  180 Minutes: Promethazine | 0 | 0
  180 Minutes: Prochlorperazine | 0 | 0
  180 Minutes: Other | 0 | 0

12. Secondary Outcome: Administration of Naloxone
Description: Yes or no, was naloxone required after the patient received the study drug?
Time Frame: 15 minutes after administration of study drug then again at 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes and at 180 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
Participants
  Yes | 0 | 0
  No | 3 | 1

13. Secondary Outcome: Change in Disposition
Description: Yes or no, did the patients disposition change as a consequence of administration of the study drug? Example would be an adverse outcome resulting in hospitalization or other escalation of care.
Time Frame: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
Participants
  Yes | 0 | 0
  No | 3 | 1

14. Secondary Outcome: Missed Diagnosis
Description: Yes or no, did the patient have a new diagnosis within the next week?
Time Frame: 7 days after administration of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
Participants
  Yes | 0 | 1
  No | 3 | 0

15. Secondary Outcome: Serious Adverse Event
Description: Yes or no, did the patient suffer a serious adverse event? Defined as death, requiring or prolonging inpatient hospitalization, resulting in persistent or significant disability/incapacity, or is considered a significant medical event by the investigator based off of medical judgement.
Time Frame: 180 minutes after administration of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
Number analyzed (Participants) | 3 | 1
Participants
  Yes | 0 | 0
  No | 3 | 1

ADVERSE EVENTS:
Time Frame: Subjects were monitored for the first 180 minutes they were in the emergency department. They were followed up to 7 days later.
Arm/Group | Intravenous Lidocaine | Intravenous Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Lidocaine (N=3) | Intravenous Hydromorphone (N=1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Feeling tired (General disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No statistical analysis was done due to enrolling only 4 subjects before the trial was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT04398316/Prot_SAP_000.pdf